CLINICAL TRIAL: NCT06517576
Title: Randomized Controlled Trial Using Remote Monitoring With an Automated Patient Engagement System and a Self-Monitoring Program With Continuous Glucose Monitors to Address Health Disparities in Type 2 Diabetes
Brief Title: Using Remote Monitoring to Address Health Disparities in Type 2 Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lawndale Christian Health Center (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Chicago (Other)
Responsible Party: Principal Investigator, Andrew Wang, Population Health Director, Lawndale Christian Health Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: LCHC-ID-10; P30DK092949 (NIH)
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Remote Patient Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Remote patient monitoring and automated patient engagement system with blood glucose monitors (Experimental): Participants in this group will receive blood glucose monitors and will check their blood glucose daily with monitoring through a digital platform and provided health coaching.
  Interventions: Device: Blood glucose monitor with Digital Platform and Health Coaching
- Self-monitoring program with continuous glucose monitors (Experimental): Participants in this group will receive continuous glucose monitors and will self monitor their blood glucose measurements with support by their care team.
  Interventions: Device: Continuous glucose monitor
- Usual care group receiving standard care (Active Comparator): Participants in this group will receive standard care for diabetes.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Blood glucose monitor with Digital Platform and Health Coaching — Blood glucose monitors will be used daily to measure blood glucose measurements.
  Other Names: Bluetooth Blood Glucose Monitor; 3011065399
  Arms: Remote patient monitoring and automated patient engagement system with blood glucose monitors
Device: Continuous glucose monitor — Continuous glucose monitors will be used daily to measure blood glucose measurements.
  Other Names: Dexcom G7 Continuous Glucose Monitoring System; 3004753838
  Arms: Self-monitoring program with continuous glucose monitors
Other: Usual Care — Usual care for type 2 diabetes
  Arms: Usual care group receiving standard care

SUMMARY:
Patient populations at community health centers, specifically Black or African American and Hispanic or Latino populations with Type 2 diabetes, experience significant health disparities. In particular, they have higher rates of diabetes-related complications and other related conditions such as myocardial infarction, cerebrovascular disease, kidney failure, blindness, neuropathy, and the risk of amputation. Diabetes affects 34 million adults in the US. Achieving a target HbA1c less than 8% can be challenging through diabetes management. Patients are able to monitor their blood glucose levels with devices such as blood glucose meters or continuous glucose monitors to facilitate diabetes management and glycemic control. Past studies have demonstrated that these devices are effective in engaging patients in the improvement of diabetes management. Current advancements in remote patient monitoring and self-monitoring have been observed to be effective in facilitating improvement in diabetes outcomes. However, the effectiveness and financial feasibility of these devices delivered in conjunction with automated patient engagement systems in remote patient monitoring programs is not well understood among underinsured, underserved, and vulnerable minority populations as they face a high-cost barrier particularly with continuous glucose monitors. To better address this gap in knowledge, this pilot study will compare and examine the effectiveness of these interventions on patient outcomes with Type 2 diabetes among populations in the West Side of Chicago. Study the comparative effectiveness among patients with uncontrolled Type 2 diabetes on insulin in an intervention group using remote patient monitoring and automated patient engagement system with blood glucose monitors to a group using a self-monitoring program with continuous glucose monitors and a usual care group receiving standard care. Conduct a feasibility analysis and financial impact of these programs among an underinsured and underserved population of Black/African Americans or Hispanic/Latinos with Type 2 diabetes.

DETAILED DESCRIPTION:
This will be conducted at a Lawndale Christian Health Center, a community health center in the West Side of Chicago that serves a largely Black or African American and Hispanic or Latino population. To accomplish this objective, Aim 1 will study the impact on patients with uncontrolled Type 2 diabetes on insulin by comparing an intervention group that features remote patient monitoring with an automated patient engagement system and health coaching using blood glucose meters compared to a group that features a self-monitoring program using continuous glucose monitoring devices and a usual care group with standard care, and Aim 2 will examine the feasibility of implementing these interventions and financial impact of each treatment group at a community health center. To understand the effect of this study on health outcomes, patient level data will be examined including primary outcomes for health measurements such as HbA1c, blood glucose, BMI/weight, estimated glomerular filtration rate (eGFR), patient-reported outcomes including medication adherence, daily activities, diabetes self-management activities, and secondary outcomes for health measurements such as LDL cholesterol, systolic and diastolic blood pressures, as well as implementation outcomes such as acceptability, appropriateness, and feasibility. The costs of implementation and delivery will be examined using a budget impact analysis. This study will be essential for informing the impact on health disparities through remote monitoring with automated patient engagement compared to self-monitoring when providing care for underinsured and underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have an assigned primary care provider
* Diagnosis of Type 2 diabetes
* Medication use is insulin
* HbA1c of 8.0% or higher

Exclusion Criteria:

* Diagnosis of chronic kidney disease at Stage 4 or higher
* Diagnosis of pregnancy
* Diagnosis of behavioral health conditions including serious mental illness or severe depression in the past 6 months.
* All participants must have a smartphone that is able to access internet services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin | Baseline and at 4 Months
  HbA1c based on blood sugar attached to hemoglobin based on lab analysis of blood.
Blood Glucose | 4 Months
  Blood glucose measurements based blood glucose monitor (BGM) and continuous glucose monitor (CGMs).
Engagement with digital platform with a daily submission of blood glucose | 4 Months
  Daily blood glucose measurements from blood glucose monitor submitted to the digital platform
Implementation - Acceptability of Intervention Measure (AIM) | Baseline and at 4 Months
  Self-reported perception among patients that this service is agreeable, palatable, or satisfactory with a likert scale of disagree to agree.
Implementation - Intervention Appropriateness Measure (IAM) | Baseline and at 4 Months
  Self-reported perception among patients that this service is fit, relevant, and compatible with a likert scale of disagree to agree.
Implementation - Feasibility of Intervention Measure (FIM) | Baseline and at 4 Months
  Self-reported perception among patients that this service is successfully used or carried out within a primary care setting with a likert scale of disagree to agree.
The Diabetes Self-Management Questionnaire (DSMQ) on eating, medication, glucose monitoring, physical activity, and healthcare use | Baseline and at 4 Months
  Self-reported perception among patients of eating behavior, medication adherence, glucose monitoring, physical activity, and healthcare use with a likert scale of applies to me very much, applies to me a considerable degree, applies to some degree, and does not apply to me.

SECONDARY OUTCOMES:
Weight | Baseline and at 4 Months
  Weight in pounds
Height | Baseline and at 4 Months
  Height in inches
Estimated glomerular filtration rate | Baseline and at 4 Months
  The eGFR based on blood test.
Low-density lipoprotein Cholesterol | Baseline and at 4 Months
  The LDL cholesterol based on blood test.
Blood Pressure | Baseline and at 4 Months
  The systolic and diastolic blood pressure using blood pressure monitor.
Clinic Visit | 4 Months
  The total count of clinic visits both virtually and on-site.
Hospitalizations | 4 Months
  The total count of hospital admissions.
Costs of Implementation | 4 Months
  Total estimated costs of implementing interventions using a budget impact analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wang, Principal Investigator — Lawndale Christian Health Center
Locations (1):
- Lawndale Christian Health Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstock RS, Aleppo G, Bailey TS, Bergenstal RM, Fisher WA, Greenwood DA, Young LA. The Role of Blood Glucose Monitoring in Diabetes Management. Arlington (VA): American Diabetes Association; 2020 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK566165/ PMID 33411424
- [Background] Schmitt A, Gahr A, Hermanns N, Kulzer B, Huber J, Haak T. The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control. Health Qual Life Outcomes. 2013 Aug 13;11:138. doi: 10.1186/1477-7525-11-138. PMID 23937988
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459